CLINICAL TRIAL: NCT07050355
Title: Combining rTMS & Aerobic Exercise to Treat Depression and Improve Post-Stroke Walking (RESTORATION)
Brief Title: Combining rTMS & Aerobic Exercise to Treat Depression and Improve Post-Stroke Walking
Acronym: RESTORATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Duke University (Other)
Responsible Party: Principal Investigator, Chris Gregory, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00137804; R01HD113299 (NIH)
Record Dates: First submitted 2025-04-03; First posted 2025-07-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Depression - Major Depressive Disorder; Walking Impairment
Keywords: stroke; rehabilitation; neuromodulation; TMS; walking; exercise
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- rTMS (Active Comparator): repetitive transcranial magnetic stimulation
  Interventions: Device: rTMS
- AEx (Active Comparator): treadmill aerobic exercise
  Interventions: Behavioral: AEx
- rTMS + AEx (Experimental): combination of repetitive transcranial magnetic stimulation and treadmill aerobic exercise
  Interventions: Device: rTMS; Behavioral: AEx

INTERVENTIONS:
Device: rTMS — Subjects will undergo rTMS to the left dorsolateral prefrontal region as a treatment for depression. Treatment will be performed three times per week for 12 weeks (36 sessions) . We will use a standard resting motor threshold (rMT) determination from unaffected abductor pollicis brevis. Treatments will be delivered at the EEG coordinate for F3 (approximating the left DLPFC) and will be found using the Beam-F3 method. A total of 5000 pulses/session will be delivered at 10Hz with an intensity of 120% of rMT.
  Arms: rTMS; rTMS + AEx
Behavioral: AEx — The goal of AEx will be 20 minutes of continuous walking at an intensity of ~70% of heart rate reserve (HRR calculated via the Karvonen method). The desired intensity will be achieved by a combination of increasing treadmill speed and incline. Rest breaks will be allowed as needed during training with the goal of progressing to 20 minutes of continuous walking.
  Arms: AEx; rTMS + AEx

SUMMARY:
Investigators primary aim is to carry out a two-site, randomized, double-blind, sham-controlled, phase II trial to systematically examine the potential for aerobic exercise (AEx) to enhance the anti-depressant benefits of rTMS in individuals with post-stroke depression (PSD).

Investigators propose to determine the efficacy of combining two known anti-depressant treatments shown to be effective in non-stroke depression, aerobic exercise (AEx) and repetitive transcranial magnetic stimulation (rTMS), on post-stroke depressive symptoms. This project is based on the idea that depression negatively affects the potential for the brain to adapt in response to treatment such that rehabilitation may not produce the same changes that it does in non-depressed individuals. Investigators believe that effective treatment for PSD will result in a virtuous cycle whereby reducing depression enhances response to rehabilitation, thereby facilitating functional gains. That is, effectively treating depression will enable individuals to better recover from stroke.

DETAILED DESCRIPTION:
This project will determine whether aerobic exercise enhances the anti-depressant benefits rTMS in individuals with PSD through a two-site, prospective, randomized trial. Over a five-year period, 96 subjects (12-60 months post-stroke) will be assigned to complete 12 weeks of treatment with rTMS, treadmill AEx or both (i.e., rTMS+AEx). Treatments will take place three times per week on non-consecutive days. Assessments of depression (HAM-D17) and walking capacity (6MWT) will be performed at two-week intervals throughout treatment as well as 12- and 24-weeks following cessation of treatment, allowing determination of the efficacy (and persistence) of training on these outcomes. Secondary outcomes will include measures of community walking (steps per day) and quality of life (Stroke Impact Scale) collected pre-, mid- and post-training, as well as at the follow-up time points. Last, investigators will explore potential biomarkers of response via assessment of PAS-induced neuroplastic potential and MR imaging to identify changes in cortical grey matter thickness.

ELIGIBILITY:
Inclusion Criteria:

* age 21-70
* stroke within the past 12 to 60 months
* screen positive for probable major depressive disorder (PHQ-9 > 10) and HAM-D17 ≥ 14
* residual paresis in the lower extremity (Fugl-Meyer LE motor score <34)
* ability to walk without assistance and without an AFO at speeds ranging from 0.2-1.0 m/s
* not currently on antidepressant medications or no changes in antidepressant dosage in the last 4 weeks and clinically stable
* HAM-D17 question #9 regarding suicide <2
* provision of informed consent.

Exclusion Criteria:

* unable to ambulate at least 150 feet prior to stroke, or experienced intermittent claudication while walking
* history of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during ADL's
* history of COPD or oxygen dependence
* history of traumatic brain injury
* blindness or severe visual impairment
* history of psychosis or other Axis I disorder that is primary
* life expectancy <1 yr.
* severe arthritis or problems that limit participation in testing or training
* history of DVT or pulmonary embolism within 6 months
* uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest
* attempt of suicide in the last 2 years or suicidal risk assessed by SCID
* history of seizures or currently prescribed anti-seizure medications
* current enrollment in a trial to enhance motor recovery
* currently participating in behavioral treatment for depression
* currently exercising ≥ 2 times per week (≥20 minutes)
* contraindications to TMS
* pregnancy or other contraindications to MRI.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Severity of depressive symptoms | baseline, after 2,4,6,8,10 and 12 weeks of treatment
  The Hamilton Depression Rating Scale (HAM-D17) is the gold-standard for clinical trial outcomes and samples a broad array of depressive symptoms. Critically, the rater administering the HAM-D17 will be clinically trained and will blinded to all other aspects of the study. For this trial, depression severity will be classified as moderate (HAM-D17 = 14-19) or severe (HAM-D = 20-25) for the purpose of stratification and diagnosed upon enrollment using the Structured Clinical Interview for Depression according to the Diagnostic & Statistical Manual of Mental Disorders, 5th Edition (DSM-V).

SECONDARY OUTCOMES:
six-minute walk test | baseline, after 2,4,6,8,10 and 12 weeks of treatment
  Distance walked in 6 minutes
Step activity monitoring | baseline, after 2,4,6,8,10 and 12 weeks of treatment
  Daily step count
Stroke Impact Scale | baseline, after 2,4,6,8,10 and 12 weeks of treatment
  Assesses multiple domains of stroke recovery on a scale from 0 to 100, including strength, hand function, activities of daily living and instrumental activities of daily living, mobility, communication, emotion, memory and thinking, and participation, with higher scores representing better recovery

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University School of Medicine, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided
Unknown at this time